CLINICAL TRIAL: NCT05495399
Title: Surgery for Limited Spine Metastases Followed by Conventional Radiotherapy or Stereotactic Body Radiation Therapy
Brief Title: Post Operative RT for Limited Spine Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202204039RINA
Record Dates: First submitted 2022-08-04; First posted 2022-08-10 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Spine Metastases
Keywords: Stereotactic body radiotherapy; Spondylectomy; Separation surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spondylectomy with Conventional RT (Experimental): Spondylectomy for involved spine level followed by conventional RT 20Gy in 5 fractions
  Interventions: Procedure: Spondylectomy
- Debulking surgery with Conventional RT (Active Comparator): Debulking surgery for involved spine level followed by conventional RT 20Gy in 5 fractions
  Interventions: Procedure: Spondylectomy; Radiation: SBRT
- Debulking surgery with SBRT (Experimental): Debulking surgery for involved spine level followed by SBRT 24Gy in 12 fractions
  Interventions: Radiation: SBRT

INTERVENTIONS:
Procedure: Spondylectomy — Patient will be randomized to treated by spondylectomy or debulking surgery. Spondylectomy implied total resection of involved spine; while debulking surgery means partial resection of involved spine.
  Arms: Debulking surgery with Conventional RT; Spondylectomy with Conventional RT
Radiation: SBRT — Patient received debulking surgery will be randomized to receive SBRT or conventional RT. SBRT means high dose per fraction compared to conventional RT.
  Arms: Debulking surgery with Conventional RT; Debulking surgery with SBRT

SUMMARY:
To evaluate patients with limited spine metastases treated with total spondylectomy followed by conventional radiotherapy or debulking surgery followed by SBRT or conventional RT. The study primary endpoint is one year local control.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had pathologically proved solid cancer, with radiographic evident limited spine metastases indicative and feasible for spondylectomy or debulking surgery.
2. Patients with maximum two continuous level of spine metastases need for surgery are eligible. Patients who have other spine metastases but not necessary for surgery are allowed.
3. A preoperative gadolinium enhance MRI should be obtained up to 8 weeks before enrollment.
4. Patients aged at least 20 years old are eligible.
5. Life expectancy of ≥ 6 months.
6. ECOG performance status 0-2 (ECOG 3-4 related to cord compression can be enrolled after physician assessment)
7. No prior RT to the index spine level(s)
8. Women of childbearing potential must practice adequate contraception
9. Patients must be able to comply with the study protocol and follow-up schedules and provide study-specific informed consent.

Exclusion Criteria:

1. Patients received prior radiotherapy to the index spine level.
2. Patients who cannot receive Gadolinium enhanced MRI due to pacemaker or metal implant or who cannot receive contrast enhanced CT scan due to impaired renal function.
3. Patients who have hematological cancer or primary spine tumor will be excluded for enrolment.
4. Patients who cannot tolerate radiotherapy immobilization.
5. Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

   1. Uncontrolled active infection requiring intravenous antibiotics at the time of registration
   2. Transmural myocardial infarction ≤ 6 months prior to registration.
   3. Life-threatening uncontrolled clinically significant cardiac arrhythmias.
   4. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
   5. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
   6. Uncontrolled psychiatric disorder.
6. Pregnant or breast-feeding women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Local control | 12 months post surgery
  Number of patients with locally controlled disease of index spine after intervention

SECONDARY OUTCOMES:
Overall survival | 12 months post surgery
  Survival from treatment to death
pain control | Every 3 months up to 1 year post surgery
  using numerical pain score to assess pain
Quality of life assessment | Every 3 months up to 1 year post surgery
  EORTC QLQ-C15 PAL
Quality of life assessment | pre surgery and 1 month after surgery
  Spine Oncology Study Group Outcomes Questionnaire 2.0 (SOSGOQ 2.0)
Quality of life assessment | Every 3 months up to 1 year post surgery
  EORTC QLQ-BM22
Treatment related toxicity | Every 3 months up to 1 year post surgery
  Using Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD sharing required by other researchers will be discussed in institution